CLINICAL TRIAL: NCT04879927
Title: Routine Evaluation of the Social Determinants of Health in Oncology: User-centered Resource Coordination and Engagement
Acronym: RESOURCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nadine McCleary, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-437
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Lung Cancer; Gastrointestinal Cancer
Keywords: Breast Cancer; Lung Cancer; Gastrointestinal Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESOURCE Matching (Experimental): Participants randomized into the intervention arm will receive customized resource matching
  Interventions: Other: Resource Matching
- Usual Care (Active Comparator): Participants randomized into the control group will receive a pre-existing pamphlet detailing DFCI resources
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Resource Matching — Resource staff involved in the customized resource matching arm of the intervention will include staff from DFCI Patient Services and DFCI Financial Counseling. Financial counseling will support patients with financial resource needs. DFCI Patient Services will provide assistance for all other patient Social Determinants of Health needs.
  Arms: RESOURCE Matching
Other: Usual Care — Patients randomized to the control group will receive a pre-existing pamphlet detailing DFCI resources.
  Arms: Usual Care

SUMMARY:
The purpose of this research is to understand how screening for patient resource needs followed by customized resource matching can improve outcomes for adults with breast, lung or gastrointestinal cancer.

DETAILED DESCRIPTION:
This research study is an intervention assessment; this is the first-time investigators are examining the impact of screening for resource needs followed by customized resource matching at Dana-Farber Cancer Institute.

* The research study procedures include screening for social determinants of health (resource) needs and, depending on study group, resource matching.
* Participants will be randomized into one of two groups.

  * Usual Care or Usual Care with customized resource matching.

It is expected that about 125 participants will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be adults age 18 or older, able to consent, scheduled for a new patient consultation in DFCI BOC, TOP or GCC. To select for patients from demographic groups vulnerable to SDoH needs, two different groups will be eligible to participate.
* Group A

  * BIPOC (Black, Latinx, Native American or Pacific Islander)
  * LEP Spanish-speaking (As indicated by the EHR)
  * Low SES (from zip code with median household income <$32,000/year) OR
  * Age 70+
* Group B

  * Any one NPIQ response indicating SDoH need
  * Health literacy/numeracy, Caregiving/relationships, OR Finances

Exclusion Criteria:

- Group A and B

-- Patients not continuing care at Dana Farber Cancer Institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients Treatment Interruption | 30 Days
  Number of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)
Number of Patients Treatment Interruption | 90 Days
  Number of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)
Number of Patients Treatment Interruption | 180 Days
  Number of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)
Rate of Treatment Interruption | 00 Days
  Rate of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)
Rate of Treatment Interruption | 90 Days
  Rate of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)
Rate of Treatment Interruption | 180 Days
  Rate of interruptions to cancer treatment (defined here as treatment hold, reduction, discontinuation or ED visits/hospitalizations as indicated by the patient medical record)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine J. McCleary, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu